CLINICAL TRIAL: NCT01181505
Title: STUDY The Effect of HNF-4A G60D Variant on the In VIVO CYP2D6 Activity By Tolterodine Pharmacokinetic Study
Acronym: HNF4a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Department of Pharmacology and PharmacoGenomics Research Center, Inje University College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06-78
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2008-11

CONDITIONS: Genotype Guided(HNF4a); Healthy Subjects
Keywords: HNF4a; CYP2D6; Toterodine; Genetic polymorphism
MeSH Terms: interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolterodine (Experimental)
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Tolterodine

SUMMARY:
This study was to investigate the pharmacokinetics of tolterodine, substrate of CYP2D6 in healthy subject in relation to the presence of HNF-4A G60D variant.

DETAILED DESCRIPTION:
After a single oral administration of 2 mg tolterodine in 31 healthy subjects (6 with the heterozygous mutation of HNF-4A G60D vs 25 subjects with wild type of that whose CYP2D6 genotype and gender were matched with variant group), blood were collected for 24hrs. Assay of tolterodine and the metabolite, 5-hyroxymethyl tolterodine was conducted using LC/MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject whose HNF4a and CYP2D6 genotype ware determined

Exclusion Criteria:

* Subject whose HNF4a and CYP2D6 genotype ware not determined

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Cmax, AUC, CL, Vd, T1/2 | 24hr

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD, PhD, Principal Investigator — Inje University